CLINICAL TRIAL: NCT07221318
Title: Evaluating the Physiological and Psychological Impact of Low-Frequency Vibration Therapy: A Longitudinal Randomized Clinical Trial
Brief Title: Evaluating a Mat-Based Biometric Vibration System for Sleep and Daily Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-25-0421
Record Dates: First submitted 2025-10-24; First posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Healthy Adult Male and Female Volunteers
Keywords: whole-body vibration therapy; sleep quality; affect; mood; relaxation therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Vibration (Kinetic Wellness Mat) (Experimental): Participants use a low-frequency kinetic wellness mat at home 3-4 days/week for 3 weeks. Each day includes a 15-minute supine session on the active mat while recording heart rate variability (HRV), plus 15-minute HRV recordings before bedtime and after waking on those same days. After each session and the next morning, participants complete brief affect check-ins (Self-Assessment Manikin: valence, arousal) and log caffeine/alcohol, exercise, and medications. All participants attend pre- and post-intervention lab visits for questionnaires, resting HRV/EEG, and a brief cognitive test (Trail Making Test). Open-label; schedule matched to control.
  Interventions: Device: Low-frequency whole-body vibration mat
- Quiet Rest Control (No Intervention): Participants complete quiet supine rest at home 3-4 days/week for 3 weeks. Each day includes a 15-minute rest period without vibration while recording HRV, plus 15-minute HRV recordings before bedtime and after waking on those same days. After each session and the next morning, participants complete brief affect check-ins (Self-Assessment Manikin: valence, arousal) and log caffeine/alcohol, exercise, and medications. All participants attend pre- and post-intervention lab visits for questionnaires, resting HRV/EEG, and a brief cognitive test (Trail Making Test). Open-label; schedule matched to the experimental arm.

INTERVENTIONS:
Device: Low-frequency whole-body vibration mat — A noninvasive, horizontal mat that delivers low-frequency mechanical vibration (≈5-16 Hz; peak-to-peak amplitude ≤0.5 mm) while participants lie supine. The active arm uses the mat at home 15 min per session, 3-4 days/week for 3 weeks, preferably in the evening (2-3 h before bedtime). On intervention days, participants record HRV during the 15-min session and complete two additional 15-min HRV recordings (immediately before bedtime and after waking) to index short-term autonomic recovery. Brief affect check-ins (valence, arousal) and logs of caffeine/alcohol, exercise, and medications are completed on those days. Pre- and post-program lab visits include questionnaires plus resting HRV and EEG. The control arm follows the identical schedule without vibration. The device provides no heat or electrical stimulation.
  Arms: Active Vibration (Kinetic Wellness Mat)

SUMMARY:
The goal of this randomized clinical trial is to learn whether a low-frequency "kinetic wellness" mat (a comfortable mat that gently vibrates) can improve stress recovery, sleep quality, mood, and attention in healthy adults ages 18-45.

The main questions it aims to answer are:

* After 3 weeks, does regular use of the vibrating mat increase heart rate variability (a noninvasive marker of the body's ability to recover from stress) and improve sleep, mood, perceived stress, and anxiety compared with no mat use?
* Do patterns of resting brain activity (measured with EEG) and heart rate variability (HRV) change from before to after the program, and are those changes related to each other?

Researchers will compare two groups: an Experimental group that uses the vibrating mat at home for 3 weeks, and a Control group that does not use the mat. Participants are randomly assigned to a group.

Participants will:

* Attend two lab visits (~60 min) for questionnaires, resting heart activity (HRV) and brain activity (EEG), and a brief attention test.
* On 3-4 days per week for 3 weeks:
* Experimental group: use the vibrating mat for 15 minutes while recording HRV.
* Control group: lie quietly for 15 minutes while recording HRV.
* Both groups: record HRV for 15 minutes before bedtime and 15 minutes after waking on those same days.
* Both groups: complete quick check-ins on feelings (after sessions and the next morning) and log caffeine/alcohol, exercise, and medications.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-45 years.
* Able to provide written informed consent.
* Apparently healthy and free of unstable cardiovascular, neurological, or psychiatric conditions per screening.
* Cleared for low-to-moderate intensity whole-body vibration delivered supine/recumbent on a mat.
* Willing and able to comply with study procedures: two lab visits; 3-week home protocol (3-4 days/week); three 15-min sessions; brief affect check-ins and daily logs.
* Willing to abstain from caffeine, alcohol, and strenuous exercise for 24 hours before each lab visit and to attend visits at the same time of day.
* Able to lie supine for 15 minutes and follow instructions for the HRV device.

Exclusion Criteria:

* Implanted electronic medical devices (e.g., pacemaker, neurostimulator).
* Uncontrolled hypertension or severe vestibular disorders.
* Current substance dependence.
* Medications known to markedly affect autonomic function or sleep architecture (e.g., beta-blockers, antiarrhythmics, sedative-hypnotics, antidepressants with strong autonomic effects).
* Diagnosed neurological or psychological disorders that substantially affect emotional processing or autonomic regulation (severe psychiatric conditions).
* Prior extensive experience with vibration therapies (to minimize expectancy bias).
* Any condition judged by study staff to contraindicate vibration exposure or preclude safe participation (including inability to tolerate supine/recumbent position).
* Unwillingness to refrain from initiating new structured exercise or relaxation programs during the study period.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Resting EEG Spectral Power | From enrollment to the end of treatment at 3 weeks
  Eyes-closed 15-minute, supine resting EEG using a 24-channel Smarting Mobi system. Preprocessing: 0.5-30 Hz band-pass, ocular SSP, ±100 µV artifact rejection, common-average reference; clean data segmented into 10-s epochs. Outcome is band power in Theta (4-8 Hz), Alpha (8-13 Hz), Beta (13-30 Hz), averaged across all electrodes and epochs (units: power; may be log-transformed for analysis). Higher values indicate stronger oscillatory activity in each band. Primary analysis compares Post-Baseline change between groups.
Resting EEG Directed Connectivity | From enrollment to the end of treatment at 3 weeks
  From the same 15-minute, eyes-closed, supine EEG. Frequency-domain Granger causality computed per 10-s epoch; spectra averaged within Theta (4-8 Hz), Alpha (8-13 Hz), Beta (13-30 Hz). Connectivity summarized across all electrodes via: (a) Global directed strength (mean of all non-diagonal influences; unitless; higher = stronger overall directed connectivity); (b) Nodal inflow and outflow (sum of incoming vs. outgoing influences for each electrode; unitless; higher = stronger received/sent influence); and (c) Pairwise directed influence (value for each electrode pair; unitless). Primary analysis compares Post-Baseline change between groups, with band-specific follow-ups.
Resting vagally mediated HRV | From enrollment to the end of treatment at 3 weeks
  Heart rate variability measured during a 15-minute, eyes-closed, supine rest in the lab. Inter-beat intervals captured with Optimal HRV; processed in Kubios (artifact correction; 4 Hz resampling; files with >5% corrected beats excluded; spectral estimates with 300-s windows, 50% overlap). Outcomes reported as:
  * RMSSD (ms): Root mean square of successive differences. Higher = greater parasympathetic (vagal) activity.
  * HF power (0.15-0.40 Hz, ms²): High-frequency power. Higher = greater parasympathetic activity.
  Primary analysis compares change (Post - Baseline) between groups for each metric; an exploratory composite (mean of RMSSD and HF z-scores) may be reported to summarize parasympathetic tone.
Longitudinal HRV Response to Intervention | Session days across Weeks 1-3
  RMSSD and HF recorded (i) during the 15-min home session (vibration vs quiet rest), (ii) 15 min before bedtime, and (iii) 15 min after waking. Outcomes are trajectories and group differences over time (linear mixed-effects). Benefit onset (threshold) will be explored via segmented regression/GAM change-point. Operational definition (pre-specified exploratory): first of two consecutive session-day recordings where RMSSD exceeds each participant's Baseline median by ≥0.10 log-units (~10% increase), sustained thereafter.

SECONDARY OUTCOMES:
Sleep Quality (PSQI Global Score) | From enrollment to the end of treatment at 3 weeks
  Pittsburgh Sleep Quality Index (0-21). Higher scores = worse sleep quality. Outcome is change in global score; report also % with PSQI >5 (poor sleep), if applicable.
Perceived Stress (PSQ Total Score) | From enrollment to the end of treatment at 3 weeks
  Perceived Stress Questionnaire total (0-30). Higher scores = more perceived stress. Outcome is change in total score.
State Anxiety (6-Item STAI Short Form) | From enrollment to the end of treatment at 3 weeks
  Six-item state anxiety scale (range 6-24). Higher scores = greater current anxiety. Outcome is change in total score.
Mood States (Brunel Mood Scale) | From enrollment to the end of treatment at 3 weeks
  BRUMS subscales scored 0-16 each. Higher = more of the construct (Tension, Fatigue); higher Vigor = more energy. Outcomes are changes in each subscale.
Cognitive Test (Trail Making Test) | From enrollment to the end of treatment at 3 weeks
  Trail Making Test Part A and Part B completion times (seconds) nd error counts for each part. Errors include sequencing mistakes. Lower times and fewer errors indicate better performance. Primary metric: Change in TMT-B completion time and B-A (set-shifting cost) from Baseline to Post between groups, considering the amount of errors.

OTHER OUTCOMES:
Affective Check-ins (Self-Assessment Manikin) | From enrollment to the end of treatment at 3 weeks
  Valence and arousal rated 1-9 (single-item pictorial scales). Higher valence = more pleasant; higher arousal = more activated. Outcomes: pre-session levels and pre-session to morning change.
Adherece | From enrollment to the end of treatment at 3 weeks
  Session completion rate (% of prescribed sessions), missed-session streaks, and proportion of analyzable HRV/EEG files. Descriptive stats; between-group comparisons by t-test or Wilcoxon as appropriate.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida International University, Biscaney Bay Campus, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
We will not share individual participant data (IPD). The dataset includes high-dimensional EEG/HRV signals and time-stamped behavioral logs from a small cohort, which pose a meaningful re-identification risk even after standard de-identification. The IRB-approved consent permits use by the study team only and does not include broad data sharing. In addition, device parameter files may contain proprietary information. We will share aggregate results and analysis specifications in publications and supplements, but not raw IPD.